CLINICAL TRIAL: NCT00067652
Title: Improving Body Image in Middle Schoolers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BODYIMAGE (completed)
Record Dates: First submitted 2003-08-25; First posted 2003-08-27 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Healthy; Body Image
MeSH Terms: interventions — Educational Status

INTERVENTIONS:
Behavioral: Education and awareness about body image issues.

SUMMARY:
The focus of this study is the development of a school-based multimedia product for the prevention of body dissatisfaction and unhealthy weight control behaviors in adolescents. The program is being designed for early adolescents, age 12-14, and will include information on maturation, healthy eating and exercise, skill building modules and media literacy awareness.

ELIGIBILITY:
Adolescents will be recruited from participating schools. Participants must be between the ages of 11-14 years.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2003-04; Study Completion 2003-11

CONTACTS AND LOCATIONS:
Locations (1):
- Inflexxion, Inc., Newton, Massachusetts, United States